CLINICAL TRIAL: NCT00000884
Title: A Randomized Phase I Safety and Immunogenicity Trial of Live Recombinant Canarypox ALVAC-HIV vCP205 Delivered by Alternate Mucosal Routes in HIV-1 Uninfected Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 027; 10577 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Injections, Intramuscular; HIV-1; Immunity, Cellular; AIDS Vaccines; HIV Seronegativity; Mucous Membrane; Antibodies, Viral; Avipoxvirus; Genetic Vectors; HIV Envelope Protein gp120; Immunity, Mucosal; Rabies Vaccines; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- 1 (Experimental): Participants will undergo treatment intramuscularly
  Interventions: Biological: ALVAC-HIV MN120TMG (vCP205); Biological: ALVAC-RG Rabies Glycoprotein (vCP65)
- 2 (Experimental): Participants will undergo treatment orally
  Interventions: Biological: MN rgp120/HIV-1 and GNE8 rgp120/HIV-1; Biological: ALVAC-HIV MN120TMG (vCP205); Biological: ALVAC-RG Rabies Glycoprotein (vCP65)
- 3 (Experimental): Participants will undergo treatment intranasally
  Interventions: Biological: MN rgp120/HIV-1 and GNE8 rgp120/HIV-1; Biological: ALVAC-HIV MN120TMG (vCP205); Biological: ALVAC-RG Rabies Glycoprotein (vCP65)
- 4 (Experimental): Participants will undergo treatment intrarectally
  Interventions: Biological: MN rgp120/HIV-1 and GNE8 rgp120/HIV-1; Biological: ALVAC-HIV MN120TMG (vCP205); Biological: ALVAC-RG Rabies Glycoprotein (vCP65)
- 5 (Experimental): Participants will undergo treatment intravaginally
  Interventions: Biological: MN rgp120/HIV-1 and GNE8 rgp120/HIV-1; Biological: ALVAC-HIV MN120TMG (vCP205); Biological: ALVAC-RG Rabies Glycoprotein (vCP65)
- 6 (Experimental): Participants will undergo treatment intranasally and intramuscularly
  Interventions: Biological: MN rgp120/HIV-1 and GNE8 rgp120/HIV-1; Biological: ALVAC-HIV MN120TMG (vCP205); Biological: ALVAC-RG Rabies Glycoprotein (vCP65)
- 7 (Experimental): Participants will undergo treatment intrarectally and intramuscularly
  Interventions: Biological: MN rgp120/HIV-1 and GNE8 rgp120/HIV-1; Biological: ALVAC-HIV MN120TMG (vCP205); Biological: ALVAC-RG Rabies Glycoprotein (vCP65)

INTERVENTIONS:
Biological: MN rgp120/HIV-1 and GNE8 rgp120/HIV-1 — Dosage will vary based on route of administration
  Arms: 2; 3; 4; 5; 6; 7
Biological: ALVAC-HIV MN120TMG (vCP205) — Dosage will vary based on route of administration
Biological: ALVAC-RG Rabies Glycoprotein (vCP65) — Dosage will vary based on route of administration

SUMMARY:
To compare the safety of ALVAC-HIV vCP205 to that of ALVAC-RG vCP65 rabies glycoprotein, delivered by a variety of mucosal routes. To evaluate the antibody, humoral, and cellular immune responses resulting from ALVAC-HIV vCP205. [AS PER AMENDMENT 8/3/98: To obtain safety data on AIDSVAX B/B boosting administered by the intramuscular and intranasal routes in the context of previous immunization via alternate mucosal routes or intramuscularly with a canarypox vector expressing HIV-1 antigens (vCP205). To obtain immunogenicity data on AIDSVAX B/B boosting.] One of the earliest observations in the HIV epidemic was the demonstration of HIV infection at mucosal surfaces of cells in the genital tract. These data suggest that priming of immune defenses of viral infected cells may be an important component in the strategy of developing an effective HIV vaccine. Direct immunization of relevant mucosal surfaces with a vectored vaccine may stimulate mucosal immunity. The ALVAC-HIV vCP205 immunogen is constructed from a live recombinant canarypox vector that has a good safety profile in volunteers and should allow mucosal induction of immunity.

DETAILED DESCRIPTION:
One of the earliest observations in the HIV epidemic was the demonstration of HIV infection at mucosal surfaces of cells in the genital tract. These data suggest that priming of immune defenses of viral infected cells may be an important component in the strategy of developing an effective HIV vaccine. Direct immunization of relevant mucosal surfaces with a vectored vaccine may stimulate mucosal immunity. The ALVAC-HIV vCP205 immunogen is constructed from a live recombinant canarypox vector that has a good safety profile in volunteers and should allow mucosal induction of immunity.

This randomized, double-blind trial evaluates the safety of and immune response to vaccination with ALVAC-HIV vCP205 given at 0, 1, 3, and 6 months. Patients are randomly assigned to 1 of 7 drug administration routes as follows:

Group A: Intramuscular Group B: Oral Group C: Intranasal Group D: Intrarectal Group E: Intravaginal Group F: Intranasal/intramuscular Group G: Intrarectal/intramuscular Twelve patients are randomized to each group, 8 of whom receive experimental therapy with ALVAC-HIV vCP205 and 4 of whom receive control therapy with ALVAC-RG vCP2058 (rabies vaccine). Women are preferentially enrolled, with a goal of 60% women (minimum of 4 women per treatment arm); only women are randomized to Group E. Blinding is maintained with respect to drug assignment rather than route of administration, after randomization. NOTE: The protocol will be amended to add 2 boost vaccinations with subunit products at approximately Months 9 and 12 when a suitable boost product is identified. [AS PER AMENDMENT 8/3/98: The protocol has been modified to include 2 booster vaccinations to be administered at 9 and 12 months. Patients in Group A receive booster vaccination with ALVAC-HIV VCP205 or ALVAC-RG intranasally. Patients in Groups B through G are boosted with AIDSVAX B/B vaccine (a bivalent vaccine consisting of MN rgp120/HIV-1 antigen and GNE8 rgp120/HIV-1 antigen in alum adjuvant) or with Imovax diploid cell rabies vaccine; vaccinations for these patients are given intramuscularly.] [AS PER AMENDMENT 11/19/98: The second booster vaccination for group A will be administered at study Month 15.]

ELIGIBILITY:
Inclusion Criteria

Volunteers must have:

* Negative ELISA for HIV within 8 weeks of immunization.
* No envelope bands in Western blot for HIV-1 within 8 weeks of immunization.
* Normal history and physical examination.

Exclusion Criteria

Co-existing Condition:

Volunteers with the following conditions are excluded:

* Medical or psychiatric condition or occupational responsibilities that preclude compliance with the protocol, including recent suicidal attempt or ideation or present psychosis.
* Active syphilis (if the serology is documented to be a false positive or due to a remote [more than 6 months] treated infection, the volunteer is eligible).
* Active tuberculosis (volunteers with a positive PPD and a normal chest x-ray showing no evidence of TB and not requiring INH therapy are eligible).
* Allergy to egg products or neomycin (used to prepare ALVAC vaccines).
* Occupational or household exposure to birds (no known pathogenicity of avipox for birds).
* Episode of severe diarrhea within 1 week prior to immunization.
* Abnormal pelvic exam with evidence of sexually transmitted disease or other genital tract infection or trauma, including vaginitis, cervicitis, ecchymosis, vulvar or cervicovaginal lesions or abrasions, or chronic cervical and/or abnormal PAP smear changes.
* Recent history of rectal bleeding or repeatedly positive hemocult test (within 1 month).
* Positive for Hepatitis B surface antigen.

Volunteers with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness (in particular, chronic inflammatory disease or gastroenteritis), malignancy, or autoimmune disease.
* History of cancer unless there has been surgical excision followed by a sufficient observation period to give a reasonable assurance of cure.
* History of anaphylaxis or history of other serious adverse reactions to vaccines.
* History of serious allergic reaction to any substance, requiring hospitalization or emergent medical care (e.g., Stevens-Johnson syndrome, bronchospasm, or hypotension).

Prior Medication:

Excluded:

* Live attenuated vaccines within 60 days of study. NOTE: Medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) are not exclusionary, but should be given at least 2 weeks away from HIV immunizations.
* Experimental agents within 30 days prior to study.
* HIV-1 vaccines or placebo received in a previous HIV vaccine trial.
* Previous immunization against rabies.

Prior Treatment:

Excluded:

* Prior hysterectomy.
* Blood products or immunoglobulin in the past 6 months.

Risk Behavior:

Excluded:

Volunteers with identifiable higher-risk behavior, or whose partners have an identifiable higher-risk behavior for HIV infection as determined by screening questions designed to identify risk factors for HIV infection (i.e., AVEG Risk Groups C or D); specific exclusions include:

* history of injection drug use within the last 12 months prior to enrollment or higher-risk sexual behavior as defined by the AVEG.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Study Completion 2000-10 (Actual)

PRIMARY OUTCOMES:
To compare the safety of ALVAC-HIV vCP205 to that of ALVAC-RG vCP65 rabies glycoprotein, delivered by a variety of mucosal routes | Throughout study
To evaluate the antibody, humoral, and cellular immune responses resulting from ALVAC-HIV vCP205 | Throughout study
To obtain safety data on AIDSVAX B/B boosting administered by the intramuscular and intranasal routes in the context of previous immunization via alternate mucosal routes or intramuscularly with a canarypox vector expressing HIV-1 antigens (vCP205) | Throughout study
To obtain immunogenicity data on AIDSVAX B/B boosting | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: P Wright, Study Chair
Locations (6):
- United States (6):
  - UAB AVEG, Birmingham, Alabama
  - JHU AVEG, Baltimore, Maryland
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - Univ. of Rochester AVEG, Rochester, New York
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee
  - UW - Seattle AVEG, Seattle, Washington